CLINICAL TRIAL: NCT05876338
Title: The Effect of Nursing Interventions Based on a Symptom Management Model on Symptom Management, Fear of Recurrence, and Quality of Life in Colorectal Cancer Survivors
Brief Title: Colorectal Cancer Survivor Symptom Management
Acronym: CRCaSSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Nazli Ozturk, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KAEK-686
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer; Survivorship
Keywords: colorectal cancer survivor; symptom management model; fear of recurrence; nursing interventions; quality of life
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRCaSSM (Experimental): CRCaSSM
  Interventions: Other: CRCaSSM
- Control (No Intervention)

INTERVENTIONS:
Other: CRCaSSM — The intervention group will receive face-to-face training, giving patient education booklet and telephone counseling based on the symptom management model. After the training, it is planned to provide telephone counseling for a total of 6 times, once every 2 weeks for 3 months.
  Arms: CRCaSSM

SUMMARY:
Objective: The aim of this study was to examine the effects of nursing interventions based on the symptom management model on symptom management, fear of recurrence, and quality of life in colorectal cancer survivors.

Method: The research was planned as a randomized controlled trial. The research is planned to be carried out at Akdeniz University Hospital. It is planned to be done with 52 patients, 26 experimental and 26 control groups. The intervention group will receive face-to-face training and telephone counseling based on the symptom management model. After the training, it is planned to provide telephone counseling for a total of 6 times, once every 2 weeks for 3 months. Participant Information Form, Memorial Symptom Assessment Scale, Fear of Cancer Recurrence Inventory and European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Scale Scale will be used to collect data.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older
2. Being able to read and write
3. Being oriented to place, time, person
4. Not having a hearing problem
5. Not having a speech problem
6. Being able to use the phone
7. Primary medical diagnosis is colorectal cancer
8. Patients who have completed primary treatment for colorectal cancer and are followed up
9. Not to relapse
10. Being in remission
11. Having a Karnofsky Performance Scale of 70% and above and being followed on an outpatient basis

Exclusion Criteria:

1.Patients with cognitive problems

Exclusion Criteria from the Sample During the Research:

1. Patient's wish to leave the study
2. Continuing the outpatient follow-up of the patient in the medical oncology outpatient clinic of another institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in symptom management at week 12 | Baseline, 4th week, 8th week and 12th week
  Memorial Symptom Assessment Scale (MSAS): The Memorial Symptom Assessment Scale is a multidimensional self-report questionnaire that evaluates 32 physical and psychological symptoms according to their frequency, severity and distress/bother to the person in the past week.The total score is the average of the responses to the distress scale items and and ranges from 0 to 4 with higher values indicating greater distress experienced from symptoms.
Change from Baseline in Fear of Cancer Recurrence at week 12 | Baseline and 12th week
  Fear of Cancer Recurrence Inventory (FCRI): It consists of 42 items with seven subscales triggers, severity, psychological distress, coping strategies, functioning impairments, insight, reassurance. FCRI, is a Likert-type scale that ranges from 0 (not at all/never) to 4 (all the time/a great deal). Increasing scores received from the scale demonstrate a high level of FCR. The minimum score to be taken from the scale is 0, and the maximum score is 168.
Change from Baseline in Quality of Life Level on the EORTC QLQ-C30 Quality of Life Scale at week 12 | Baseline and 12th week
  EORTC QLQ-C30 Quality of Life Scale(European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire): This Scale was developed to measure the quality of life of patients with cancer. It includes 30 questions and three sub-dimensions: General Well-Being, Functional Difficulties, and Symptom Control. The maximum score on the scale is 100, and the minimum is 0. High scores on the functional sub-dimension indicate good/healthy functional status, high scores on the symptom sub-dimension indicate high levels of symptoms and/or problems, and high scores on the global health status/quality of life sub-dimension indicate good quality of life.
Change from Baseline in Quality of Life Level on the EORTC QLQ-CR29 Quality of Life | Baseline and 12th week
  EORTC QLQ-CR29 The QLQ-CR29 includes 29 items that evaluate symptoms (gastrointestinal, urinary, pain and others) and functional areas (sexual, body image and others). Similar to the EORTC QLQ-C30, the QLQ-CR29 has a Likert scale of four response categories (item 48 requires a yes or no answer). All patient-rated scores are linearly converted into a scale from 0 to 100 for both the QLQ-C30 and QLQ-CR29.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Arikan, Study Director — Akdeniz University
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No